CLINICAL TRIAL: NCT04266288
Title: Rapid Antidepressant Response to Ketamine and Impact on Healthcare Utilization After Administration in the Emergency Department
Brief Title: Effectiveness of Ketamine for Depression and Suicidal Ideation in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MercyOne Des Moines Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Bress, PharmD, Pharmacist, MercyOne Des Moines Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMC2019-46
Record Dates: First submitted 2020-02-04; First posted 2020-02-12 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Depression; Depression Severe; Depression Acute; Depression and Suicide; Suicidal Ideation
Keywords: Ketamine; Depression; Suicidal Ideation; Emergency Department
MeSH Terms: conditions — Depression; Suicide; Suicidal Ideation; Emergencies | interventions — Ketamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Ketamine 0.5 mg/kg in 0.9% sodium chloride, total volume 50 mL via intravenous infusion over 40 minutes for one dose.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): 0.9% sodium chloride, total volume 50 mL via intravenous infusion over 40 minutes for one dose
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Ketamine — Active drug
  Other Names: Ketalar
  Arms: Ketamine
Drug: Sodium Chloride 0.9% — Placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of a low-dose ketamine infusion on depression symptoms within the Emergency Department (ED) visit, and healthcare utilization after leaving the ED, when administered in the ED for depression or suicidal ideation.

DETAILED DESCRIPTION:
Patients will be identified based on either a chief complaint of suicidal ideation, suicide attempt, or severe depression, or if the patient indicates during intake assessment that they have thoughts of harming or killing their self. Identified patients will be assessed by the ED provider for inclusion and exclusion criteria. If the patient is a candidate for the trial and gives their informed consent for enrollment, they will be randomized to receive either ketamine or placebo by a computer program that maintains blinding. The patient will be assessed by psychiatry for disposition and treatment plan prior to receiving the study drug, and will be reassessed four hours after the infusion. Thirty days after the patient leaves the hospital (either leaves from the ED or is discharged from inpatient admission), they will be contacted to follow up on their healthcare utilization after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Presenting to the ED with a chief complaint of severe depression or suicidality, or presenting to the ED with any other chief complaint but answering "yes" to "Thoughts of harming/killing yourself?" during intake/triage

Exclusion Criteria:

* Acute mania or psychosis
* Enrollment in trial during a prior emergency department visit
* History of ketamine abuse or dependence
* Known hypersensitivity to ketamine
* Acute intoxication with any drug of abuse (including alcohol)
* Pregnancy or lactation
* Any condition that would place the patient at serious risk of harm from an increase in blood pressure (e.g. history of intracerebral hemorrhage, aneurysmal vascular disease, or arteriovenous malformation)
* Assessing provider does not want to enroll patient for any other reason, based on their clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Depression Symptom Response | Baseline, 4 hours
  Patients will be classified as a responder or non-responder, with a response defined as a decrease by 50% or greater for the combined depressive symptom scores of the Brief Psychiatric Rating Scale (BPRS), which includes the following domains: emotional withdrawal, guilt feelings, depressed mood, blunted affect, feelings of inferiority, and suicidal ideation. The total depressive symptom score ranges from 6-42, with a higher score indicating a higher level of severity. Response rate will be compared between the treatment and placebo groups.
ED Return Visit | 30 days from discharge
  Number of return visits to the emergency department for any psychiatric reason

SECONDARY OUTCOMES:
Outpatient follow-up | 30 days from discharge
  Patients will be contacted at 30 days from discharge to obtain outpatient follow-up data. The two results for this outcome are "yes" or "no" to having at least one outpatient visit, either with a psychiatry provider or with a primary care provider to obtain psychiatric care. The number of outpatient visits an individual patient reports, if greater than one, does not affect this outcome. Attempts will be made to confirm each reported visit with the provider to minimize the potential for subject bias.
Intoxication | Baseline, 2 hours, 4 hours
  Change in Visual Analog Scale for Intoxication (VAS-High), which ranges from 0 to 8, with a higher score indicating a greater level of impairment.
Changes in Individual Psychiatric Symptoms | Baseline, 4 hours
  Change in Brief Psychiatric Rating Scale (BPRS) individual symptom scores, with each range from 1-7, with a higher score indicating a higher level of severity. There are 18 total symptoms evaluated on the BPRS.
Length of stay | Time from arrival in ED to discharge, either directly from the ED or after inpatient admission. Average length of stay is less than 14 days.
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Bress, PharmD, Principal Investigator — MercyOne Des Moines Medical Center; Adnan Iqbal, MD, Principal Investigator — MercyOne Des Moines Medical Center
Locations (1):
- MercyOne Des Moines Medical Center, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No